CLINICAL TRIAL: NCT06777030
Title: Role of Exosomes in Pancreatic Cancer Progression
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: EXOPanc
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of tumour tissue, blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present pilot study is set up with the objective of identifying circulating markers in the biological fluids (blood and urine) of subjects with pancreatic carcinoma and their association with disease stage, to evaluate their potential use as predictive and diagnostic markers for this tumor of difficult early diagnosis and often inauspicious prognosis.

DETAILED DESCRIPTION:
The study is cross-sectional, single-center, spontaneous, in human tissues. It is a pilot study to gather evidence on the content of extracellular vesicles/exosomes in patients with pancreatic cancer.

The study will be performed on tumor tissue, blood and urine samples. Tissue will be obtained by needle biopsy (fine needle biopsy - FNB) during echoendoscopic examination.

The study aims to characterize the content of extracellular vesicles/exosomes in the biological fluids of subjects with pancreatic cancer with the goal of identifying new markers for this disease. To this end, the following will be carried out:

* an ex vivo and in vitro characterization study of the secretion of these extracellular vesicles/exosomes with analysis of their contents in terms of proteins and nucleic acids;
* a study of the mechanisms of epithelial-mesenchymal transition (EMT), invasion and aggressiveness to highlight a possible association between the secretion of these vesicles and the oncological stage of pancreatic carcinoma;

ELIGIBILITY:
Inclusion criteria:

* People with pancreatic cancer
* 18 years old
* Obtaining informed consent.

Exclusion criteria:

* Patients who do not need or cannot perform endoscopy with biopsy sampling;
* patients with a previous or active neoplastic pathology, different from pancreatic neoplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves the enrollment of patients hospitalized for diagnostic-therapeutic evaluation of pancreatic neoformation. In particular, patients will be included for whom biopsy sampling of the pancreatic lesion by means of an ultrasound-guided needle biopsy is planned during hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Characterise the extracellular vesicle/exosome content of patients with pancreatic carcinoma. | At baseline, visit V1.
  The study aims to characterize the extracellular vesicles/exosomes content in the biological fluids of subjects suffering from pancreatic carcinoma with the aim of identifying new markers for this disease. To this end, the following will be carried out:
  * a study of ex vivo and in vitro characterisation of the secretion of these extracellular vesicles/exosomes with analysis of their content in terms of proteins and nucleic acids;
  * a study of mesenchymal epithelium transition (EMT), invasion and aggression mechanisms to highlight a possible association between secretion of these vesicles and the oncological stage of pancreatic carcinoma;

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Henry Umberto Eusebi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided